CLINICAL TRIAL: NCT00802555
Title: A Phase 1b Safety Study of ARQ 197 in Cirrhotic Patients With Hepatocellular Carcinoma (HCC)
Brief Title: Safety Study of ARQ 197 in Cirrhotic Patients With Hepatocellular Carcinoma (HCC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ArQule, Inc., a subsidiary of Merck Sharp & Dohme LLC, a subsidiary of Merck & Co., Inc. (Rahway, NJ USA) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARQ 197-114
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: Cirrhosis; Hepatocellular Carcinoma
Keywords: HCC; Cirrhotic Patients with Hepatocellular Carcinoma
MeSH Terms: conditions — Fibrosis; Carcinoma, Hepatocellular | interventions — ARQ 197

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ARQ 197 (Experimental)
  Interventions: Drug: ARQ 197

INTERVENTIONS:
Drug: ARQ 197 — 360 mg administered twice daily until disease progression, unacceptable toxicity, or other discontinuation criterion is met

SUMMARY:
Multi-center, single-arm Phase 1b study designed to evaluate safety and tolerability of ARQ 197 in cirrhotic patients with HCC.

DETAILED DESCRIPTION:
Study designed to evaluate safety and tolerability of ARQ 197 in cirrhotic patients with HCC who have received ≤2 prior systemic regimens for HCC, and whose liver disease severity is categorized as Class A and B per Child-Pugh Classification.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent granted prior to initiation of any study-specific screening procedures, given with the understanding that the patient has the right to withdraw from the study at any time, without prejudice
* 18 year of age or older
* Histologically or cytologically confirmed HCC (not required if: a hepatic lesion is >2cm in diameter , is suggestive of HCC at radiology and α-fetoprotein (AFP) is > 200 mg/mL)
* Barcelona Clinic Liver Cancer (BCLC) staging Category27 A, B or C that can not benefit from treatments of established efficacy and/or higher priority
* Cirrhotic status of Child-Pugh Class A and B without ascites or with slight ascites that can be recognized only by imaging techniques and/or managed easily with diuretics (e.g. 100 mg spironolactone per day and/or furosemide 40 mg/day)
* Cirrhotic status confirmed by one of the following methods/evidence:
* Biopsy
* Endoscopy showing gastrointestinal tract varices
* Evidence of portal hypertension on imaging studies such as dilated portal vein, collateral circulation
* ECOG PS ≤1
* Not more than two prior systemic regimens for HCC and the last treatment must have been completed ≥4 weeks prior to first dose of ARQ 197
* Local or loco-regional therapy (i.e., surgery, radiation therapy, hepatic arterial embolization, chemoembolization, radiofrequency ablation, percutaneous ethanol injection, or cryoablation) must have been completed ≥4 weeks prior to first dose of ARQ 197
* Measurable disease as defined by revised Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1. Tumor lesions selected as target lesion(s) at baseline should not have been previously treated with local therapy (naïve tumor lesion)
* Adequate bone marrow, liver, and renal functions, defined as:
* Platelet count ≥ 60 × 10^9/L
* Hemoglobin ≥ 8.5 g/dL
* Absolute neutrophil count (ANC) ≥1.5 × 10^9/L
* Total bilirubin ≤ 3 mg/dL
* Alanine transaminase (ALT) and aspartate transaminase (AST) ≤ 5 × upper limit of normal (ULN)
* Serum creatinine ≤1.5 × ULN
* International normalized ratio (INR) ≤ 2.3 or PT ≤ 6.0 seconds above control. Patients who are therapeutically anticoagulated with an agent such as coumadin or heparin are allowed to participate provided that no prior evidence of underlying abnormality exists in these parameters
* Albumin ≥ 2.8 g/dL
* Women of childbearing potential must have a negative pregnancy test performed within seven days prior to the start of study drug
* Male and female subjects of child-bearing potential must agree to use double-barrier contraceptive measures, oral contraception, or avoidance of intercourse during the study and for 90 days after last investigational drug dose received

Exclusion Criteria:

* Previous or concurrent cancer that is distinct from HCC in primary site or histology, EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta, Tis & T1). Any cancer curatively treated >3 years prior to enrollment is permitted
* History of cardiac disease: congestive heart failure defined as Class II to IV per New York Heart Association (NYHA) classification; active coronary artery disease (CAD); previously diagnosed bradycardia or other cardiac arrhythmia, or uncontrolled hypertension; myocardial infarction occurred within 6 months prior to study entry (myocardial infarction occurred > 6 months prior to study entry is permitted)
* Active clinically serious infections defined as ≥ Grade 2 according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 3.0
* Substance abuse, medical, psychological or social conditions that may, in the opinion of the Investigator, interfere with the patient's participation in the study or evaluation of the study results
* Any condition that is unstable or which could jeopardize the safety of the patient and his/her protocol compliance
* Known HIV (human immunodeficiency virus) infection
* Pregnancy or breast-feeding
* History of liver transplant
* Inability to swallow oral medications
* Clinically significant gastrointestinal bleeding occurring ≤4 weeks prior to first dose of ARQ 197

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of ARQ 197 when administered in cirrhotic patients diagnosed with HCC

SECONDARY OUTCOMES:
To evaluate time to disease progression (TTP), objective response rate (ORR), and disease control rate (DCR) in patients with HCC
To evaluate dynamic changes of hepatocyte growth factor (HGF), vascular endothelial growth factor (VEGF), and soluble c-Met in patients' peripheral blood that are associated with ARQ 197 treatment

CONTACTS AND LOCATIONS:
Locations (5):
- United States (2):
  - Dallas, Texas
  - Houston, Texas
- Italy (2):
  - Bologna
  - Milan
- Barcelona, Spain